CLINICAL TRIAL: NCT06913374
Title: Dicycle Versus Tri-cycle High-dose Dexamethasone in Adult ITP: a Multicenter Randomized Controlled Trial
Brief Title: The Study of Different Cycles of High-dose Dexamethasone in the Treatment of ITP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX 2v3 in ITP
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Thrombocytopenia
Keywords: ITP; Dexamethasone
MeSH Terms: conditions — Thrombocytopenia | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group DEX2 (Experimental): In group DEX2, dexamethasone was administered orally at 40 mg per day for two cycles (days1-4, and days 11-14).
  Interventions: Drug: Dexamethasone
- group DEX3 (Experimental): In group DEX3, dexamethasone was administered orally at 40 mg per day for three cycles (days1-4, days 11-14, and days 21-24).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — given orally at 40 mg per day for two cycles (days1-4, and days 11-14).
  Other Names: DEX
  Arms: group DEX2
Drug: Dexamethasone — given orally at 40 mg per day for three cycles (days1-4, days 11-14, and days 21-24).
  Other Names: DEX
  Arms: group DEX3

SUMMARY:
Primary immune thrombocytopenia is an autoimmune disorder characterised by decreased platelet counts and increased bleeding risk. Corticosteroids have been the standard initial treatment of primary immune thrombocytopenia for more than 30 years. The aim of this randomized controlled trial is to compare the efficacy and safety of high-dose dexamethasone in treating new-diagnosed primary immune thrombocytopenia (ITP) in di-cycle and tri-cycle.

DETAILED DESCRIPTION:
In this multicentre, open-label, randomized controlled trial, about 118 new-diagnosed ITP patients will be enrolled from five tertiary medical centres in China. Eligible participants are randomly assigned (1:1) to 2 groups: group DEX2 and group DEX3. In group DEX2, dexamethasone was administered orally at 40 mg per day for two cycles (days1-4, and days 11-14). In group DEX3, dexamethasone was administered orally at 40 mg per day for three cycles (days1-4, days 11-14, and days 21-24). The clinical effect, onset time, duration of efficacy and adverse reactions were observed to compare the efficacy and safety of two different plans.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of the screening.
* Participant may be male or female.
* Participant has a confirmed diagnosis of newly diagnosed ITP according to the 2019 International Working Group assessment at screening, and has a baseline platelet count of less than 30 × 10^9 cells per L or had bleeding manifestations, or both.

Exclusion Criteria:

* Participant has evidence of a secondary cause of immune thrombocytopenia (e.g. leukemia, lymphoma, common variable immune- deficiency, systemic lupus erythematosus, autoimmune thyroid disease, past medical history of untreated H. pylori infection) or to drug treatments (e.g. heparin, quinine, antimicrobials, anticonvulsants) or participant has a multiple immune cytopenia, e.g. Evan's syndrome.
* Participant has clinically life-threatening bleeding (e.g. central nervous system bleeding, menorrhagia with significant drop in hemoglobin).
* Participant has a history of coagulopathy disorders other than ITP.
* Participant has a history of arterial or venous thromboembolism (e.g. stroke, transient ischemic attach, myocardial infarction, deep vein thrombosis or pulmonary embolism) within the 6 months prior to randomization or requires anticoagulant treatment.
* Participant has 12-lead ECG with changes considered to be clinically significant upon medical review at baseline.
* Participant has severe renal impairment (glomerular filtration rate less than 45ml/min/1.73 m2).
* Participant has 3 × upper limit of normal of any of the following: alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase.
* Participant with any of the following conditions: severe immunodeficiency, active or previous malignancy, human immunodeficiency virus (HIV), hepatitis B or C virus infection, pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response | Month 6
  Sustained response was defined as platelet count maintained above 30 × 10^9/L with an absence of bleeding symptoms or no requirement for additional ITP treatment for six consecutive months following achievement of initial response. Complete response was defined as a platelet count of 100 × 10^9 cells per L or higher and an absence of bleeding. Partial response was defined as a platelet count of 30×10^9 cells per L or higher, but less than 100×10^9 cells per L, and at least a doubling of the baseline platelet count and an absence of bleeding.

SECONDARY OUTCOMES:
Initial response | Day 24
  Initial responses were assessed by day 24. Complete response was defined as a platelet count of 100 × 10^9 cells per L or higher and an absence of bleeding. Partial response was defined as a platelet count of 30×10^9 cells per L or higher, but less than 100×10^9 cells per L, and at least a doubling of the baseline platelet count and an absence of bleeding.
Time to response | 24 days
  Time to response was defined as the time from treatment initiation to achieve a complete response or a partial response, whichever came first, assessed up to day 24.
Duration of response | 12 months
  Duration of response was defined as the time from achievement of a complete response or a partial response to the loss of response (platelet count <30 × 10^9 cells per L; measured on two occasions more than 1 day apart or the presence of bleeding).
Bleeding scores | 12 months
  Bleeding symptoms were graded according a standardized bleeding scale specific to primary immune thrombocytopenia on the basis of site and severity of bleeding by Khellaf et al (PMID: 15951296). A modification was made to exclude age from the original scale so that only bleeding symptoms were described. At each visit, we recorded bleeding scores.Scores ranged from 0 to 59, with higher values indicating higher bleeding risk.
Health-related quality of life assessment | 12 weeks
  Health-related quality of life was assessed using a self-administered immune thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) at baseline and at week 12. Scores ranged from 0 to 100, with higher values indicating better quality of life.
The number of participants with Adverse events | 12 months
  Adverse events were graded according to the Common Terminology Criteria for Adverse Events (version 4.0). At each visit, we recorded adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong university, Jinan, Shandong, China